CLINICAL TRIAL: NCT07295548
Title: Postoperative Management of Patients Undergoing Head and Neck Microvascular Free Flap Reconstructive Surgery: is Admission to an Intensive Care Unit Necessary?
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Simone Mauramati, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: RIA_COMPL
Record Dates: First submitted 2025-12-03; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Reconstructive Surgery; Head and Neck Microvascular Free Flap

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU (Intensive Care Unit) Cohort
  Interventions: Procedure: free flap surgery
- non-ICU (Intensive Care Unit) Cohort
  Interventions: Procedure: free flap surgery

INTERVENTIONS:
Procedure: free flap surgery — evaluation of major and minor complications, flap failure rates and length of hospital stay in patients undergoing free flap surgery admitted to intensive care unit and in those admitted to an Otolaryngology specialty ward

SUMMARY:
The aim of our study is to assess if patients undergoing head and neck free flap reconstructive surgery admitted to the ICU have equivalent postoperative outcomes to those admitted to an Otolaryngology specialty ward

DETAILED DESCRIPTION:
Reconstruction with microvascular free flaps has become the standard of care for various surgical defects in head and neck region. Free flap reconstructive surgery is considered a major surgery with long intraoperative time and critical post-operative care. Close monitoring of the flap viability is of utmost importance especially in the first 48-72 hours after surgery, during which most of the vascular complications could occur; this interval is also critical for eventual successful salvage of an ischemic flap. Despite the delicacy of the matter worldwide there's not yet consensus about which is the most appropriate protocol for postoperative management after free flap surgery. Many patients undergoing free flap surgery are initially admitted to intensive care unit (ICU), even in cases of patients that do not meet any specific indication supporting the need for admission to an ICU setting. There are several reasons to this behaviour but, unfortunately, a post-operative stay in ICU is associated with increased nosocomial infections, complications and costs. The primary aim of this study will be to assess safety and postoperative outcomes (major and minor complications, flap failure rates and length of hospital stay) of patients undergoing reconstructive surgery with microvascular free flaps admitted to ICU compared to a non-ICU ward.The primary objective is to identify in which group of patients minor complications are more frequently encountered (complications that do not require surgical treatment in the operating room are considered as minor).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing Head and Neck oncological demolitive surgery and reconstruction using free or pedicled flaps at the Fondazione IRCCS Policlinico San Matteo, Pavia

Exclusion Criteria:

* patients treated for Head and Neck cancer without flap reconstruction (e.g., only chemotherapy-radiotherapy, only radiotherapy, only immunotherapy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing Head and Neck oncological demolitive surgery and reconstruction using free or pedicled flaps at the Fondazione IRCCS Policlinico San Matteo, Pavia
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-10-13 (Estimated); Study Completion 2027-10-13 (Estimated)

PRIMARY OUTCOMES:
difference in proportions of minor complications in the two groups of patients | up to 24 months
  the difference in proportions of minor complications in the two groups of patients (ICU compared to a nonICU ward)

SECONDARY OUTCOMES:
difference in proportions of major complications and necrosis in the two groups of patients | up to 24 months
  the difference in proportions of major complications and necrosis in the two groups of patients (ICU compared to a nonICU ward).
difference in length of hospitalisation in the two groups of patients | up to 24 months
  the difference in length of hospitalisation in the two groups of patients (ICU compared to a non ICU ward)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy